CLINICAL TRIAL: NCT04404673
Title: Multicenter Prospective Evaluation of Urinary and Sexual Dysfunctions After Rectal Cancer Resection
Brief Title: Urinary and Sexual Dysfunctions Evaluation After Rectal Resection
Acronym: EURECA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Other Study IDs: 2987
Record Dates: First submitted 2020-05-19; First posted 2020-05-27 (Actual); Last update posted 2020-05-27 (Actual); Status verified 2020-05

CONDITIONS: Rectal Cancer
Keywords: Urinary dysfunction; Sexual dysfunction; Rectal surgery; Minimally invasive surgery
MeSH Terms: conditions — Rectal Neoplasms; Sexual Dysfunction, Physiological

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Open rectal resection
  Interventions: Procedure: Evaluation of urinary and sexual dysfunction after rectal resection
- Laparoscopic rectal resection
  Interventions: Procedure: Evaluation of urinary and sexual dysfunction after rectal resection
- Robotic rectal resection
  Interventions: Procedure: Evaluation of urinary and sexual dysfunction after rectal resection
- Trans-anal TME (Ta-TME)
  Interventions: Procedure: Evaluation of urinary and sexual dysfunction after rectal resection

INTERVENTIONS:
Procedure: Evaluation of urinary and sexual dysfunction after rectal resection — Comparison among the 4 different surgical approaches for urinary and sexual function

SUMMARY:
Advances in the treatment of rectal cancer over the past two decades have improved survival and significantly reduced surgery-related morbidity. As a result, post-treatment quality of life (QoL) issues have become increasingly important. Urinary and sexual functions can be significantly altered after rectal resection, mainly due to the iatrogenic lesions of the pelvic autonomous lexus. Of note, their incidence is reported up to 70% and 30%, respectively. Despite the importance of this topic, most of the studies present in the literature are difficult to interpret for a variety of reasons. Firstly, both sexual and urinary dysfunctions lack a standardized definition. Secondly, the absence of baseline data, missing data, small sample sizes, and heterogeneity in the use of validated and nonvalidated instruments are the main limitation in drawing conclusive results. As additional factor, no clear evidence is present in the literature regarding the best approach to be used in order to preserve as much as possible both the sexual and urinary functionalities and to guarantee, at the same time, an adequate and oncologically correct rectal resection. Moreover, no data are currently present regarding the impact of pre-operative chemo-radiotherapy on the urinary and sexual functionalities. The main objective of the investigator's prospective study will be to define in a subjective manner which technique (open, laparoscopic, robot-assisted and Ta-TME) will guarantee the best urinary and sexual outcomes after rectal resection (with or without pre-operative chemo-radiotherapy) for the treatment of rectal carcinomas.

Thus, the primary endpoint will the post-operative evaluation at 1, 6 months and 1 year of the urinary and sexual functions by means of specific questionnaires.

Secondary endpoints will be:

* to investigate which technique (open, robotic, laparoscopic and trans-anal total mesorectal excision (TaTME)) more favorably correlate with urinary and sexual functions after radiochemotherapy (NAD+);
* the comparison of both the urinary and sexual dysfunction incidence on the base of the distance of the rectal tumor from the anal verge and the evaluation of the best approach to be used (open, laparoscopic, TaTME or robot-assisted) in relation to the tumor height;
* the short- (postoperative morbidity and histopathological data) and long-term (overall and disease-free survival) outcomes comparison among the open, laparoscopic, TaTME and robotic rectal resection.

ELIGIBILITY:
Inclusion Criteria:

* All patients with a histopathological proven diagnosis of rectal carcinoma undergoing curative surgical resection

Exclusion Criteria:

* Patients aged < 18 years
* Inability to give informed consent
* Emergent surgeries
* Previous prostatic and/or colorectal surgery for benign or malignant diseases
* Preoperative sexual disorders (Female Sexual Function Index, FSFI ≤ 26.55 ; International Index Erectile Function , IIEF < 16)
* International Consultation on Incontinence Questionnaire > 5
* Clinically evident Benign Prostatic Hypertrophy (BPH) (International Prostatic Symptoms Score, IPSS > 20)
* Preoperative diagnosis of fecal and/or urinary incontinence.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with a diagnosis of rectal cancer referred to one of the centers involved in the study during the study period
Sampling Method: Non-Probability Sample
Enrollment: 1172 (Estimated)
Dates: Start 2020-02-21 (Actual); Primary Completion 2024-02-20 (Estimated); Study Completion 2024-02-20 (Estimated)

PRIMARY OUTCOMES:
Urinary and sexual outcomes after rectal resection | At 1 month after surgery
  Which technique (open, laparoscopic, robot-assisted and Ta-TME) will guarantee the best urinary and sexual outcomes after rectal resection (with or without pre-operative chemo-radiotherapy) for the treatment of rectal carcinomas
Urinary and sexual outcomes after rectal resection | At 6 months after surgery
  Which technique (open, laparoscopic, robot-assisted and Ta-TME) will guarantee the best urinary and sexual outcomes after rectal resection (with or without pre-operative chemo-radiotherapy) for the treatment of rectal carcinomas
Urinary and sexual outcomes after rectal resection | At 12 months after surgery
  Which technique (open, laparoscopic, robot-assisted and Ta-TME) will guarantee the best urinary and sexual outcomes after rectal resection (with or without pre-operative chemo-radiotherapy) for the treatment of rectal carcinomas

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione Policlinico Universitario Agostino Gemelli IRCCS di Roma, Rome, Lazio, Italy

IPD SHARING:
Plan to Share IPD: Undecided